CLINICAL TRIAL: NCT03663985
Title: FALCOn (Facteur AnthropoLogique Cancer Orl) Evaluation Des Facteurs Anthropologiques, Socio-culturels et Psychologiques Des Praticiens Qui Conditionnent la Prise de décision Pour Les Patients Atteints de Cancer Des VADS
Brief Title: FALCOn (Facteur AnthropoLogique Cancer Orl)
Acronym: FALCOn
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Onco-Occitanie (Toulouse) (Unknown); University Hospital, Caen (Other); Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 17HLSHS01
Record Dates: First submitted 2018-07-20; First posted 2018-09-10 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Cancer; Head and Neck Carcinoma
Keywords: head and neck squamous cell carcinoma; surgery; anthropology; sociology
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Groupe FALCOn — The objective of the study is to determine what are the anthropo-sociological factors in the surgeon, the oncologists and radiotherapists influencing decision making in ENT carcinology.

SUMMARY:
There are no studies on practitioner-related factors influencing decision-making in the field of carcinology of aerodigestive carcinomas. The objective of the study is to determine what are the anthropo-sociological factors in the surgeon, the oncologists and radiotherapists influencing decision making in ear, nose, and throat carcinology. Special attention will be paid to the practitioner's gender, age, geographical origin, place and institution of training, place of practice, volume of patients treated, access to or without reconstruction by microsurgery, his tendency or aversion to risk taking.

* Main objectives : To determine the individual professional and non-professional characteristics influencing physicians' decision-making in oncology of aerodigestive carcinomas between choices:

  1. Surgery
  2. Radio and / or chemotherapy
  3. Support care
  4. Neo-adjuvant chemotherapy and reassessment
* Secondary objectives : Identify if certain patient profiles may lead to heterogeneous treatment decisions i.e. Human Papillomavirus status, age, comorbidities, autonomy, etc.

DETAILED DESCRIPTION:
Actually, there are no studies on practitioner-related factors influencing decision-making in the field of carcinology of aerodigestive carcinomas.

The objective of the study is to determine what are the anthropo-sociological factors in the surgeon, the oncologists and radiotherapists influencing decision making in ear, nose, and throat carcinology.

Special attention will be paid to the practitioner's gender, age, geographical origin, place and institution of training, place of practice, volume of patients treated, access to or without reconstruction by microsurgery, his tendency or aversion to risk taking.

This questionnaire will include the items age, sex, place and date of obtaining a medical degree, whether or not obtaining the specialization in cancer, profession of surgeon / oncologist / radiotherapist, place of practice with type of institution (University hospital, Private clinic, etc.) volume of patients treated per year, access or not to reconstructions by microsurgery. The answers to the questionnaire will be anonymous.

Practitioners' attitudes towards risk and uncertainty will be evaluated by 4 validated tools in behavioral science:

1. Self-assessment of attitude towards risk in different areas (Likert scale)
2. Monetary choice when earnings probabilities are known (attitude to risk)
3. Monetary choice when earnings probabilities are not known (attitude towards uncertainty)
4. Experience of Allais Seven clinical cases will serve as a basis for the creation of clinical vignettes.

A standard case will be part of these vignettes allowing a validation on the respect of the guidelines. The other 6 clinical cases will be cleavants and 36 vignettes will be created by crossing the 6 previous clinical cases with 6 different patient profiles on their social and demographic characteristics (age, comorbidity, sex, isolation)

The experimental plan will take the form of a Latin Square to propose (in addition to the standard case), 6 vignettes to each practitioner by ensuring that all the factors will be presented in a balanced and random way.

In a first phase, the online questionnaire including the vignettes will be evaluated within the sponsor center and by two ear, nose, and throat surgeons from two other centers who have agreed to participate in the project in order to verify its feasibility before global sending.

ELIGIBILITY:
Inclusion Criteria:

* Ear, nose and throat surgeons, oncologists specializing in oncology of aerodigestive carcinomas, radiation therapists specialized in oncology of aerodigestive carcinomas exercising in France

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Aerodigestive carcinomas surgeons, oncologists specializing in oncology of aerodigestive carcinomas, radiation therapists specialized in oncology of VADS exercising in France. Email addresses accessible via GETTEC / GORTEC / GERCOR / SFORL / UNICANCER.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the anthropological, socio-cultural and psychological factors of the practitioners which condition the decision making for the patients with aero-digestive carcinomas. | 2018, September to December
  An analysis using a classification method will define a typology of therapeutic choices given their aggression and potential risk.
  These typologies of prescriptions will then be confronted with the characteristics of physicians in terms of propensity for risk taking and their socio-demographic characteristics using a chi2 test (univariate) and a logistic regression (or polynomial if a binary typology cannot be released (multivariate).
  Variability of choice and influence of physician characteristics on these choices will also be analyzed based on patient characteristics
  Expected results :
  * Impact of socio-professional characteristics on the decision-making in oncology of aerodigestive carcinomas.
  * Impact of psychological factors ie tendency to take risk

SECONDARY OUTCOMES:
Determination of clinical recommendations choices of the health practitioners for different clinical cases of aerodigestive carcinomas | 2018, September to December
  7 clinical cases will serve as a basis for the creation of clinical vignettes: A standard case (T2N1M0 pelvi-lingual carcinoma, good general condition patient) will be part of these vignettes allowing a validation on the respect of the guidelines.The other 6 clinical cases will be cleavants.
  The experimental plan will take the form of a Latin Square to propose (in addition to the standard case), 6 vignettes to each practitioner by ensuring that all the factors will be presented in a balanced and random way.
  Practitioners will be asked to give their clinical recommendations for each clinical case presented.
Self assessment of willingness to take risk (by health practitioners themselves) | 2018, September to December
  All the health practitioners will be asked to self-evaluate their propensity to take risk using a 11-point Likert scale ranging from "not at all willing to take risks" to "fully prepared to take risks" in 4 different domains including their daily life, their personal finances, their patient's health and their own health. The Likert scale used in this test is a 0-10 scale where 0 means "not at all willing to take risks" and 10 means "fully prepared to take risks"
Evaluation of health practitioners' risk attitude | 2018, September to December
  Individual attitudes toward risk will be obtained through certainty equivalent elicitation of a lottery. Using a scrollbar, respondents will be asked to provide the amount of money that makes them indifferent between gaining it for sure or playing the lottery giving them 500 euros with half a chance and nothing otherwise. The expected gain of this lottery is 250 euros, so when the elicited certainty equivalent is inferior (equal/superior) to 250 euros, the respondent is considered as risk averse (neutral/seeking).
Evaluation of health practitioners' uncertainty attitude | 2018, September to December
  Individual attitudes towards uncertainty will be obtained through certainty equivalent elicitation of a lottery where the probability of gain is unknown. Using the same scrollbar, respondents will be asked to provide the amount of money that makes them indifferent between gaining it for sure or playing the lottery giving them 500 euros with an unknown probability and nothing with an unknown probability.
Evaluation of health practitioners' rationality attitude | 2018, September to December
  Individual rationality attitudes will be obtained through an Allais test. The expected utility theory is an axiomatic model of decision under uncertainty and is often considered as a normative model of rationality. Allais and Kahneman and Tversky proposed a set of two binary choices that allow to test the independence axiom of the expected utility theory under risk and therefore the adequacy of an individual to the model.
  The Allais task will be assessed with this 2 questions:
  Choice 1: Which option do you prefer?
  * Option A gives you 100% of chance to win 2000$
  * Option B gives you 80% of chance to win 3000$ and 20% of chance to win 0$ Choice 2: Which option do you prefer?
  * Option C which gives you 25% of chance to win 2000$ and 75% of chance to win 0$
  * Option D which gives you 20% of chance to win 3000$ and 80% of chance to win 0$ Choice pattern AD indicates a violation of rationality. Same line of reasoning applies for the choice pattern BC.

CONTACTS AND LOCATIONS:
Overall Officials: Agnès DUPRET-BORIES, PhD, Principal Investigator — Institut Claudius Regaud
Locations (1):
- Institut Claudius Regaud, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Krahenmann-Muller S, Virgini VS, Blum MR, da Costa BR, Collet TH, Martin Y, Cornuz J, Zimmerli L, Gaspoz JM, Bauer DC, Kerr EA, Aujesky D, Rodondi N. Patient and physician gender concordance in preventive care in university primary care settings. Prev Med. 2014 Oct;67:242-7. doi: 10.1016/j.ypmed.2014.08.004. Epub 2014 Aug 10. PMID 25117521
- [Result] Andersen MR, Urban N. Physician gender and screening: do patient differences account for differences in mammography use? Women Health. 1997;26(1):29-39. doi: 10.1300/J013v26n01_03. PMID 9311098
- [Result] Franks P, Clancy CM. Physician gender bias in clinical decisionmaking: screening for cancer in primary care. Med Care. 1993 Mar;31(3):213-8. doi: 10.1097/00005650-199303000-00003. PMID 8450679
- [Result] Frank E, Harvey LK. Prevention advice rates of women and men physicians. Arch Fam Med. 1996 Apr;5(4):215-9. doi: 10.1001/archfami.5.4.215. PMID 8769910
- [Result] Arrington AK, Jarosek SL, Virnig BA, Habermann EB, Tuttle TM. Patient and surgeon characteristics associated with increased use of contralateral prophylactic mastectomy in patients with breast cancer. Ann Surg Oncol. 2009 Oct;16(10):2697-704. doi: 10.1245/s10434-009-0641-z. Epub 2009 Aug 4. PMID 19653045
- [Result] Tsugawa Y, Jena AB, Figueroa JF, Orav EJ, Blumenthal DM, Jha AK. Comparison of Hospital Mortality and Readmission Rates for Medicare Patients Treated by Male vs Female Physicians. JAMA Intern Med. 2017 Feb 1;177(2):206-213. doi: 10.1001/jamainternmed.2016.7875. PMID 27992617
- [Result] Mehrotra A, Reid RO, Adams JL, Friedberg MW, McGlynn EA, Hussey PS. Physicians with the least experience have higher cost profiles than do physicians with the most experience. Health Aff (Millwood). 2012 Nov;31(11):2453-63. doi: 10.1377/hlthaff.2011.0252. PMID 23129676
- [Result] Meier P, Duvernoy CS. Influence of gender of physicians and patients on guideline-recommended treatment of chronic heart failure in a cross-sectional study. Eur J Heart Fail. 2009 Jun;11(6):631; author reply 631-2. doi: 10.1093/eurjhf/hfp056. Epub 2009 Apr 27. No abstract available. PMID 19398490
- [Result] Berthold HK, Gouni-Berthold I, Bestehorn KP, Bohm M, Krone W. Physician gender is associated with the quality of type 2 diabetes care. J Intern Med. 2008 Oct;264(4):340-50. doi: 10.1111/j.1365-2796.2008.01967.x. Epub 2008 Apr 4. PMID 18397244
- [Result] Reid RO, Friedberg MW, Adams JL, McGlynn EA, Mehrotra A. Associations between physician characteristics and quality of care. Arch Intern Med. 2010 Sep 13;170(16):1442-9. doi: 10.1001/archinternmed.2010.307. PMID 20837830
- [Result] Schieber AC, Delpierre C, Lepage B, Afrite A, Pascal J, Cases C, Lombrail P, Lang T, Kelly-Irving M; INTERMEDE group. Do gender differences affect the doctor-patient interaction during consultations in general practice? Results from the INTERMEDE study. Fam Pract. 2014 Dec;31(6):706-13. doi: 10.1093/fampra/cmu057. Epub 2014 Sep 11. PMID 25214508
- [Result] Allais, M. (1953). L'extension des théories de l'équilibre économique général et du rendement social au cas du risque. Econometrica, Journal of the Econometric Society, 269-290.
- [Derived] Chabrillac E, Lamy S, Grosclaude P, Cros F, Vairel B, Sarini J, Vergez S, Nebout A, Bories P, Dupret-Bories A. The impact of physician's characteristics on decision-making inhead and neck oncology: Results of a national survey. Oral Oncol. 2022 Jun;129:105895. doi: 10.1016/j.oraloncology.2022.105895. Epub 2022 Apr 29. PMID 35500434